CLINICAL TRIAL: NCT06108856
Title: Effect of Dialysis Adequacy in Nutritional Status and Quality of Life in Hemodialysis Patients
Brief Title: Dialysis Adequacy in Nutritional Status in Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, George san dawoud bebawy, Principal Investigator, Cairo University
Other Study IDs: dialysis adequacy
Record Dates: First submitted 2023-09-27; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Dialysis Adequacy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Hemodialysis machine — machine by which people undergo dialysis on it.

SUMMARY:
Assess nutrition status in hemodialysis patients and effect adequacy of hemodialysis on it.

Effect of dialysis adequacy and nutritional status in patients' quality of life.

DETAILED DESCRIPTION:
Patients with end-stage renal disease (ESRD) are unable to sustain life without hemodialysis. So, adequacy of hemodialysis is the main treatment for this patient.

Adequacy of hemodialysis can be appeared on patient clinically by improve Quality of life and life expectancy, increase appetite and weight gain, control blood pressure, no bone disease, control of acidosis and anemia, Relief of uremic symptoms as nausea, vomiting, fatigue, anorexia, weight loss, muscle cramps, pruritus, or changes in mental status.

Malnutrition is a major issue in patients undergoing hemodialysis and is observed in approximately 20% - 70% of this group. Malnutrition is a serious predictive factor for mortality and morbidity accompanied by an increase in the rate of hospitalization, less physical activity, lower quality of life.

An imbalance between energy and protein gain and food metabolism, metabolic acidosis, dietary restrictions, anorexia and poor appetite, protein and nutrient loss during dialysis, underlying diseases, such as cardiovascular problems, infection, poor nutrition management, inadequate dialysis, etc. are among influencing factors on the nutrition of hemodialysis patients.

Among patients undergoing hemodialysis, 6% to 8% suffer from severe malnutrition and 30% - 65% from mild malnutrition. The results of some studies have shown that one of the important causes of malnutrition is low dialysis adequacy in patients undergoing hemodialysis.

Malnutrition is associated with an increase in morbidity, a decrease in functional capacity, and a greater number and duration of hospital admissions, all of which may cause a low health-related quality of life (QOL) and impact patients' emotional, physical, and psychosocial health.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in regular haemodialysis .
2. patients above 18 years

Exclusion Criteria:

1. Patients with thyroid illness.
2. Patients with acute infection.
3. Patients with major surgeries.
4. Patients with malignancy.
5. Patients with liver cirrhosis.
6. patient with inflammatory bowel diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient on regular hemodialysis above 18 years without acute infection, major surgeries, recent trauma, or liver cirrhosis.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Effect of dialysis adequacy in nutritional status in haemodialysis patients by Body mass index (BMI) and Anthropometric measurements. | baseline
  assess how dialysis adequacy affect nutritional status using :
  1. Body mass index (BMI) : calculated based on the weight (kg)/height (m2) formula as it divide into :
     1. underweight (BMI < 18.5) worse outcome
     2. normal weight (BMI from 18.5 to 25) better outcome .
     3. overweight (BMI = 25 - 30).
     4. obese (BMI >30) .
        b)Anthropometric measurements :
     <!-- -->
     1. weight in kilograms .
     2. height in meters.
     3. waist circumference in centimeters.
     4. hip circumference in centimeters.
     5. mid arm circumference in centimeters.

REFERENCES:
- [Background] Kutsal DA, Kursat S, Inci A, Ulman C, OzanUtuk I. The relationship between malnutrition subgroups and volume parameters in pre-dialysis patients. Saudi J Kidney Dis Transpl. 2016 Jan;27(1):81-7. doi: 10.4103/1319-2442.174082. PMID 26787571
- [Background] Chan M, Kelly J, Batterham M, Tapsell L. Malnutrition (subjective global assessment) scores and serum albumin levels, but not body mass index values, at initiation of dialysis are independent predictors of mortality: a 10-year clinical cohort study. J Ren Nutr. 2012 Nov;22(6):547-57. doi: 10.1053/j.jrn.2011.11.002. Epub 2012 Mar 9. PMID 22406122